CLINICAL TRIAL: NCT03467438
Title: Efficacy of Zinc L-carnosine (Hepilor®) in Maintaining Remission of Gastroesophageal Reflux Disease: a Randomised, Double-blind, Placebo-controlled Study
Brief Title: Efficacy of Zinc L-carnosine in Maintaining Remission of Gastroesophageal Reflux Disease
Acronym: GERDILOR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Antonio Di Sabatino, Head of the First Department of Internal Medicine, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GERDILOR17
Record Dates: First submitted 2018-03-05; First posted 2018-03-16 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: heartburn; pyrosis; regurgitation
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn | interventions — polaprezinc

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The manufacturer will provide packages of the investigational medical product/placebo that are indistinguishable. Every package have a code written on it; only the manufacturer knows whether that code refers to the IMD or placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Experimental): Zinc-l-carnosine, liquid oral formulation, 75mg twice daily (20mL, using the measuring cup, twice daily), to be swallowed on an empty stomach (waiting at least one hour from the last meal).
  Interventions: Drug: Zinc-l-carnosine
- B (Placebo Comparator): Placebo, liquid oral formulation, 75mg twice daily (20mL, using the measuring cup, twice daily), to be swallowed on an empty stomach (waiting at least one hour from the last meal).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Zinc-l-carnosine — Patients will be asked to take the investigational product as already mentioned (blindly).
  Arms: A
Other: Placebo — Patients will be asked to take placebo as already mentioned (blindly).
  Arms: B

SUMMARY:
Gastroesophageal reflux disease (GERD), according to the Montreal classification, is defined as a condition that develops when the reflux of stomach contents causes troublesome symptoms and/or complications. GERD, as clinically defined by the presence of heartburn, acid regurgitation, or both, at least once a week, is a global disease, being one of the most common gastroenterological disorders worldwide that affects roughly 10-30% of the general population in the Western world and less than 10% of the Asian populations. GERD complications may be life threatening and range from reflux esophagitis to Barrett's oesophagus and, eventually, adenocarcinoma.

Zinc L-carnosine (brand name in Italy: Hepilor®) is a chelate compound of zinc and L-carnosine, with a long history of more than 20 years of clinical use in Japan that has recently become available in Italy for the treatment of any condition that requires a mucosal protection and mucosal repair within the gastrointestinal tract, thus including GERD. However, clinical data in western countries are limited. The aim of this double-blind, placebo-controlled study is to demonstrate the efficacy of Zinc-l-carnosine in maintaining GERD clinical remission during a 12-week treatment.

DETAILED DESCRIPTION:
The investigators hypothesise that Zinc-l-carnosine is able to maintain GERD remission, thus improving the quality of life of these patients. A comparison with a placebo is necessary, as GERD symptoms may be heavily influenced by the nocebo/placebo effect.

This is a post-marketing, single center, double-blind, and randomized, placebo-controlled, parallel study. Patients with GERD treated with an 8-week cours of proton pump inhibitors will be randomize and receive either Zinc-l-carnosine or placebo for 12-week. GERD symptoms will be assessed with a questionnaire (modified GERD questionnaire by Locke) monthly for 12 weeks and after a 4-week wash-out. Also, quality of life will be assessed at baseline and at 12 weeks with the 36-item short form survey (SF-36).

ELIGIBILITY:
Inclusion Criteria:

* written informed consent to participate
* be male or female patients ≥ 18 years old, with an established diagnosis of GERD
* have a diagnosis of GERD that is established clinically in case of typical symptoms (heartburn and acid regurgitation ≥ once weekly) or with 24-hour esophageal impedence monitoring in case of atypical symptoms not responsive to proton pump inhibitors (PPIs) or in case of unclear diagnosis
* have been treated with an 8-week course of PPI (as per gold-standard treatment of GERD) before entering the study

Exclusion Criteria:

* any medical condition that requires chronic therapy with PPIs or H2 antagonists; anti-acid agents must be discontinued within the study period
* oesophageal motility disorders
* allergy or intolerance to Hepilor® (it contains parahydroxybenzoate that may cause allergies)

  * inconclusive diagnosis of GERD and related symptoms
  * patients with active H. pylori infection (diagnosed with any of the available tests)
  * previous major oesophageal surgery
  * history of any advanced/relevant organ dysfunction, in particular chronic kidney disease, chronic liver disease of any aetiology, hearth failure
  * any concomitant medical condition with a poor prognosis (< 3 months)
  * pregnant females
  * inability to conform to the protocol
  * treatment with any investigational drug within the previous 3 months
  * any subject not able to express/understand the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-11-22 (Actual); Primary Completion 2020-04-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Gastroesophageal reflux disease (GERD) remission | 4 weeks
  GERD remission will be assessed according to the modified GERD questionnaire by Locke et al. GERD remission is established if any mild symptom does not occur 2 or more days a week, or if any moderate/severe symptom does not occur more than one day a week.
Gastroesophageal reflux disease (GERD) remission | 8 weeks
  GERD remission will be assessed according to the modified GERD questionnaire by Locke et al. GERD remission is established if any mild symptom does not occur 2 or more days a week, or if any moderate/severe symptom does not occur more than one day a week.
Gastroesophageal reflux disease (GERD) remission | 12 weeks
  GERD remission will be assessed according to the modified GERD questionnaire by Locke et al. GERD remission is established if any mild symptom does not occur 2 or more days a week, or if any moderate/severe symptom does not occur more than one day a week.

SECONDARY OUTCOMES:
36 item short form health survey | 12 weeks
  Quality of life will be assessed with SF-36 at baseline and after 12 weeks of treatment. The difference between the two groups will be compared at the end of treatment.
Sustained GERD remission | 16 weeks
  GERD remission will be assessed according to the modified GERD questionnaire by Locke et al. after a 4-week wash-out (week 16). GERD remission is established if any mild symptom does not occur 2 or more days a week, or if any moderate/severe symptom does not occur more than one day a week.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Italy

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD), anonymized and aggregated, that underlie results in a publication.
Supporting Information: SAP, CSR
Time Frame: Only on future articles that will be published.

REFERENCES:
- [Background] Vakil N, van Zanten SV, Kahrilas P, Dent J, Jones R; Global Consensus Group. The Montreal definition and classification of gastroesophageal reflux disease: a global evidence-based consensus. Am J Gastroenterol. 2006 Aug;101(8):1900-20; quiz 1943. doi: 10.1111/j.1572-0241.2006.00630.x. PMID 16928254
- [Background] Arakawa T, Satoh H, Nakamura A, Nebiki H, Fukuda T, Sakuma H, Nakamura H, Ishikawa M, Seiki M, Kobayashi K. Effects of zinc L-carnosine on gastric mucosal and cell damage caused by ethanol in rats. Correlation with endogenous prostaglandin E2. Dig Dis Sci. 1990 May;35(5):559-66. doi: 10.1007/BF01540402. PMID 2331952
- [Background] Locke GR 3rd, Talley NJ, Fett SL, Zinsmeister AR, Melton LJ 3rd. Prevalence and clinical spectrum of gastroesophageal reflux: a population-based study in Olmsted County, Minnesota. Gastroenterology. 1997 May;112(5):1448-56. doi: 10.1016/s0016-5085(97)70025-8. PMID 9136821
- [Background] Locke GR, Talley NJ, Weaver AL, Zinsmeister AR. A new questionnaire for gastroesophageal reflux disease. Mayo Clin Proc. 1994 Jun;69(6):539-47. doi: 10.1016/s0025-6196(12)62245-9. PMID 8189759